CLINICAL TRIAL: NCT06272929
Title: Serum Elafin: A Biomarker in Behcet Disease and Its Relation to Vascular Involvement and Disease Activity
Brief Title: Serum Elafin and Vascular Affection in Behcet Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lobna Amer Araby Ahmed, Assiut, Assiut University
Other Study IDs: behcet and vascular
Record Dates: First submitted 2024-02-16; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Behcet Disease and Vascular Affection
MeSH Terms: conditions — Behcet Syndrome | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 45 patients with behcet disease
  Interventions: Device: doppler ultrasound
- 45 healthy participants
  Interventions: Device: doppler ultrasound

INTERVENTIONS:
Device: doppler ultrasound — doppler US

SUMMARY:
To measure the level of serum elafin in patients with BD. To assess the relation between serum elafin levels and disease activity. To evaluate the vascular complications in BD and determine their relationship with disease activity.

To assess the correlation between serum elafin and vascular affection and their relation with disease activity.

DETAILED DESCRIPTION:
Behçet's disease (BD) is a chronic, multisystemic, inflammatory disease characterized by recurrent oral and genital ulcers and multiple systemic involvements. Elafin is a serine protease inhibitor produced mainly by epithelial cells. Its expression is upregulated by proinflammatory cytokines such as IL-1β and TNF-α that are potent stimulants of neutrophil activation, it counteracts the destructive effects of neutrophil elastase .Interestingly, previous reports documented the role of serum elafin in the pathogenesis of BD.In fact, vascular complications may be one of the earliest manifestations leading to the diagnosis of BD. There is no reliable tool to identify vascular wall inflammation in BD, except for detecting intravascular thrombosis with ultrasonography (US). Previous studies investigated arterial vessel wall thickness with US (mostly in carotid arteries) in BD . Venous wall inflammation presents with deep vein thrombosis and superficial thrombophlebitis . It was stated that lower extremity vein wall thickness (VWTs)was increased in BD patients independently of vascular activity and important in the diagnosis . However, studies in the literature evaluated only lower extremity VWTs, whereas the relationship of VWT with disease activity has not been emphasized .

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed as BD. Age of all participants (20-45) years.

Exclusion Criteria:

Age <20 or >45 years. Other autoimmune diseases. Cardiovascular diseases (heart failure, myocardial ischemia). Possible related risk factors (e.g. diabetes, dyslipidemia, smoking). chronic conditions (e.g. chronic kidney disease, malignancy, autoimmune diseases).

Ages: 20 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Patients diagnosed as BD. Age of all participants (20-45) years.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Measuring the level of serum Elafin in patients with BD in comparison to healthy participants. | within one year
  Measuring the level of serum Elafin in patients with BD in comparison to healthy participants.

REFERENCES:
- [Background] Calamia KT, Schirmer M, Melikoglu M. Major vessel involvement in Behcet's disease: an update. Curr Opin Rheumatol. 2011 Jan;23(1):24-31. doi: 10.1097/BOR.0b013e3283410088. PMID 21124084
- [Background] Kutlay A, Kose AA. Serum Elafin as a Potential Marker of Disease Activity in Behcet's Disease. Indian J Dermatol. 2023 Jul-Aug;68(4):372-376. doi: 10.4103/ijd.ijd_913_22. PMID 37822392
- [Background] Yazici Y, Hatemi G, Bodaghi B, Cheon JH, Suzuki N, Ambrose N, Yazici H. Behcet syndrome. Nat Rev Dis Primers. 2021 Sep 16;7(1):67. doi: 10.1038/s41572-021-00301-1. PMID 34531393